CLINICAL TRIAL: NCT01523392
Title: A Randomized, Open-Label, Multiple Dose, Crossover, Multiple Center Study of the Antiplatelet Effects of Ticagrelor Versus Clopidogrel in African American Patients With Stable Coronary Artery Disease
Brief Title: A Pharmacodynamic Study With Ticagrelor in African American Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5130L00013
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-09

CONDITIONS: Stable Coronary Artery Disease
Keywords: Stable Coronary Artery Disease, CAD
MeSH Terms: interventions — Ticagrelor; Clopidogrel

ARMS (2):
- Ticagrelor (Experimental)
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Min - 90mg/Max - 180mg tablets (loading dose)
  Arms: Ticagrelor
Drug: Clopidogrel — 75mg (once daily)/Max - 600mg tablets (loading dose)
  Arms: Clopidogrel

SUMMARY:
The purpose of this study is to assess the pharmacodynamic effect of ticagrelor in African American patients with stable coronary artery disease.

DETAILED DESCRIPTION:
A Randomized, Open-Label, Multiple Dose, Crossover, Multiple Center Study of the Antiplatelet Effects of Ticagrelor versus Clopidogrel in African American Patients with Stable Coronary Artery Disease

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent before initiation of any study-related procedures
* Male or female patients aged 18 years or older
* Documented stable CAD fulfilling and taking 75-100mg ASA daily treatment
* Females must be post menopausal or surgically sterile Self-identified as African American

Exclusion Criteria:

* Any indication for oral anticoagulant (e.g., atrial fibrillation, mitral stenosis or prosthetic heart valve) or dual antiplatelet treatment (e.g., clopidogrel, prasugrel, ASA dose other than 75 to 100 mg daily) during study period
* Patients who had ACS or stent placed within 12 months of screening Patients with a history of moderate or severe hepatic impairment
* Current smokers, including the use of tobacco containing products in the past 1 month of randomization Patients required dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Carlson, MD, Study Director — AstraZeneca Pharmaceuticals Room C3B-718PO Box 15437 Wilmington, DE 19850-5437 USA
Locations (8):
- United States (8):
  - Research Site, Newark, Delaware
  - Research Site, Wilmington, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Towson, Maryland
  - Research Site, Beaumont, Texas

REFERENCES:
- [Derived] Waksman R, Maya J, Angiolillo DJ, Carlson GF, Teng R, Caplan RJ, Ferdinand KC. Ticagrelor Versus Clopidogrel in Black Patients With Stable Coronary Artery Disease: Prospective, Randomized, Open-Label, Multiple-Dose, Crossover Pilot Study. Circ Cardiovasc Interv. 2015 Jul;8(7):e002232. doi: 10.1161/CIRCINTERVENTIONS.114.002232. PMID 26152562
- See also: D5130L00013_Study_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=485&filename=D5130L00013_Study_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from 8 participating centers in the United States from 28 March 2012 until 04 September 2013
Pre-assignment Details: 50 patients screened; 34 patients randomized; 30 patients completed the study (7, 8, or 9 days of both treatments), and 31 completed follow-up
Groups:
- Ticagrelor (Period 1) Then Clopidogrel (Period 2) Sequence: Ticagrelor 180 milligrams (mg) loading dose followed by 90 mg twice daily (bd) for 7, 8 or 9 days (Period 1), and then clopidogrel 600 mg loading dose followed by 75 mg once daily (od) for 7, 8 or 9 days (Period 2)
- Clopidogrel (Period 1) Then Ticagrelor (Period 2) Sequence: Clopidogrel 600 mg loading dose followed by 75 mg od for 7, 8 or 9 days (Period 1), and then ticagrelor 180 mg loading dose followed by 90 mg bd for 7, 8 or 9 days (Period 2)
Period: Treatment Period 1
Arm/Group | Ticagrelor (Period 1) Then Clopidogrel (Period 2) Sequence | Clopidogrel (Period 1) Then Ticagrelor (Period 2) Sequence
Started | 20 | 14
Completed | 17 | 14
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Did not complete 7-9 days of treatment. | 1 | 0
Period: Washout Period - 10 to 14 Days
Arm/Group | Ticagrelor (Period 1) Then Clopidogrel (Period 2) Sequence | Clopidogrel (Period 1) Then Ticagrelor (Period 2) Sequence
Started | 18 (1 patient did not complete 7-9 days of Period 1 treatment but continued in the Washout and Period 2) | 14
Completed | 17 | 14
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Treatment Period 2
Arm/Group | Ticagrelor (Period 1) Then Clopidogrel (Period 2) Sequence | Clopidogrel (Period 1) Then Ticagrelor (Period 2) Sequence
Started | 17 | 14
Completed | 17 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Analysis Set for demography (N=34) - included all patients who signed informed consent and were randomized into the study.
Groups:
- Ticagrelor (Period 1) Then Clopidogrel (Period 2) Sequence: Ticagrelor 180 mg loading dose followed by 90 mg bd for 7, 8 or 9 days (Period 1), and then clopidogrel 600 mg loading dose followed by 75 mg od for 7, 8 or 9 days (Period 2)
- Total: Total of all reporting groups
Arm/Group | Ticagrelor (Period 1) Then Clopidogrel (Period 2) Sequence | Clopidogrel (Period 1) Then Ticagrelor (Period 2) Sequence | Total
Number analyzed (Participants) | 20 | 14 | 34
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0
  >=18 to <65 years | 12 | 10 | 22
  >= 65 years | 8 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 12 | 11 | 23
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 20 | 14 | 34
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 20 | 14 | 34
Region of Enrollment [Number; unit: Participants]
  United States | 20 | 14 | 34

OUTCOME MEASURES:

1. Primary Outcome: Inhibition of the P2Y12 Receptor as Measured by Platelet Reaction Unit (PRU) From VerifyNow™ (a Platelet Function Test Developed by Accumetrics) at 2 Hours After Loading Dose
Time Frame: At 2 hours after the loading dose
Population: Pharmacodynamic (PD) Analysis Set (N=32) - included all participants for whom PD data was available with no major protocol deviations thought to significantly affect the PD of ticagrelor or clopidogrel
Measure: Least Squares Mean (95% Confidence Interval); unit: PRU
Groups:
- Ticagrelor: Ticagrelor 180 mg loading dose followed by 90 mg bd for 7, 8 or 9 days
- Clopidogrel: Clopidogrel 600 mg loading dose followed by 75 mg od for 7, 8 or 9 days
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 29 | 28
PRU | 27.6 [4.9 to 50.2] | 211.2 [188.3 to 234.0]
Statistical Analysis 1: Comparison: Ticagrelor vs Clopidogrel; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Model contained treatment group, period, and sequence as fixed effects and a random effect for patient within sequence; Mean Difference (Final Values) = -183.6, 95% CI 2-sided [-213.9 to -153.3], Standard Error of Mean 14.68 — Ticagrelor minus clopidogrel

2. Secondary Outcome: Inhibition of the P2Y12 Receptor as Measured by PRU From VerifyNow™ at 0.5 Hour and 8 Hours After Loading Dose
Time Frame: At 0.5 hour and 8 hours after the loading dose
Population: PD Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: PRU
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 29 | 28
PRU
  0.5 hours | 166.3 [137.9 to 194.8] | 270.1 [241.3 to 298.8]
  8 hours (N=28 ticagrelor, N=27 clopidogrel) | 27.2 [4.3 to 50.2] | 192.6 [169.3 to 215.8]
Statistical Analysis 1: Comparison: Ticagrelor vs Clopidogrel; Analysis at 0.5 hours after loading dose; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Model contained treatment group, period, and sequence as fixed effects, and a random effect for participant within sequence; Mean Difference (Final Values) = -103.8, 95% CI 2-sided [-142.5 to -65.0], Standard Error of Mean 18.79 — Ticagrelor minus clopidogrel
Statistical Analysis 2: Comparison: Ticagrelor vs Clopidogrel; Analysis at 8 hours after loading dose; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -165.3, 95% CI 2-sided [-197.4 to -133.3], Standard Error of Mean 15.45 — Ticagrelor minus clopidogrel

3. Secondary Outcome: Inhibition of the P2Y12 Receptor as Measured by PRU From VerifyNow™ at 2 Hours and 8 Hours on Day 7 After Multiple Doses and at End of Dosing Interval on Day 8
Time Frame: At 2 hours and 8 hours on Day 7 after multiple doses and at end of dosing interval on Day 8
Population: PD Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: PRU
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 28 | 27
PRU
  2 hours on Day 7 (N=27 for clopidogrel) | 22.9 [1.4 to 44.4] | 157.8 [135.9 to 179.8]
  8 hours on Day 7 | 28.5 [7.7 to 49.2] | 146.5 [125.6 to 167.4]
  End of dosing interval on Day 8 | 39.3 [17.8 to 60.7] | 172.7 [151.2 to 194.2]
Statistical Analysis 1: Comparison: Ticagrelor vs Clopidogrel; Analysis at 2 hours on Day 7 after multiple doses; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -135.0, 95% CI 2-sided [-160.4 to -109.5], Standard Error of Mean 12.35 — Ticagrelor minus clopidogrel
Statistical Analysis 2: Comparison: Ticagrelor vs Clopidogrel; Analysis at 8 hours on Day 7 after multiple doses; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -118.1, 95% CI 2-sided [-143.9 to -92.2], Standard Error of Mean 12.55 — Ticagrelor minus clopidogrel
Statistical Analysis 3: Comparison: Ticagrelor vs Clopidogrel; Analysis at end of dosing interval on Day 8; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -133.4, 95% CI 2-sided [-159.7 to -107.1], Standard Error of Mean 12.77 — Ticagrelor minus clopidogrel

4. Secondary Outcome: Ticagrelor Plasma Concentrations After the Loading and Maintenance Doses
Description: The standard deviation (SD) is the geometric SD
Time Frame: Predose, 0.5 hour, 2 hours, 8 hours from loading dose; 0, 2 hours, 8 hours and 12 hours from last dose
Population: Pharmacokinetic (PK) Analysis Set - included all patients for whom at least one valid PK reading was available
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- Ticagrelor (Treatment Period 1); Ticagrelor (Treatment Period 2): Ticagrelor 180 mg loading dose followed by 90 mg bd for 7, 8 or 9 days
Arm/Group | Ticagrelor (Treatment Period 1) | Ticagrelor (Treatment Period 2)
Number analyzed (Participants) | 20 | 11
ng/mL
  Baseline (0 pre-dose hours) | 1.0 (1.0) | 1.2 (1.8)
  0.5 hours after the loading dose | 206.6 (5.2) | 33.7 (8.2)
  2 hours after the loading dose | 1167.3 (1.8) | 756.9 (1.9)
  8 hours after the loading dose - Period 1 N=19 | 395.9 (1.5) | 141.9 (12.1)
  0 hours after multiple doses - Period 1 N=18 | 168.4 (7.3) | 187.4 (2.1)
  2 hours after multiple doses - Period 1 N=18 | 324.6 (8.9) | 608.8 (1.9)
  8 hours after multiple doses - Period 1 N=18 | 179.2 (7.4) | 311.3 (1.7)
  End of dosing interval on Day 8 - Period 1 N=18 | 284.9 (2.2) | 295.7 (1.9)

5. Secondary Outcome: AR-C124910XX (an Active Metabolite of Ticagrelor) Plasma Concentrations After the Loading and Maintenance Doses
Description: The standard deviation (SD) is the geometric SD
Time Frame: Predose, 0.5 hour, 2 hours, 8 hours from loading dose and 0, 2 hours, 8 hours and 12 hours from last dose
Population: Pharmacokinetic (PK) Analysis Set - included all patients for whom at least one valid PK reading was available
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ticagrelor (Treatment Period 1) | Ticagrelor (Treatment Period 2)
Number analyzed (Participants) | 20 | 11
ng/mL
  Baseline (0 pre-dose hours) | 1.0 (1.0) | 1.0 (1.0)
  0.5 hours after the loading dose | 9.8 (4.9) | 2.3 (3.2)
  2 hours after the loading dose | 222.6 (2.7) | 150.9 (2.5)
  8 hours after the loading dose - Period 1 N=19 | 119.0 (1.7) | 54.8 (7.5)
  0 hours after multiple doses - Period 1 N=18 | 93.2 (5.8) | 74.5 (2.0)
  2 hours after multiple doses - Period 1 N=18 | 136.7 (6.3) | 172.3 (1.7)
  8 hours after multiple doses - Period 1 N=18 | 89.8 (5.6) | 112.6 (1.3)
  End of dosing interval on Day 8 - Period 1 N=18 | 140.8 (1.9) | 110.3 (1.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signature of the informed consent throughout the treatment period including the follow up visit (approximately 11 weeks for each participant).
Description: Adverse events were solicited at each scheduled visit and could be reported by the participant at any time during the study. When summarizing Treatment Period 1 and Treatment Period 2 totals, each participant was counted only once for an individual adverse event, regardless of whether it occurred on ticagrelor, clopidogrel or both.
Arm/Group | Ticagrelor | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/31
Other Adverse Events (participants affected / at risk) | 5/34 | 2/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=34) | Clopidogrel (N=31)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) — Occurred 14 days after the last dose of ticagrelor
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ticagrelor (N=34) | Clopidogrel (N=31)
Haemorroidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Application site bruise (General disorders) | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Vaginal haemmorhage (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AstraZeneca (AZ) for review at least 60 days in advance of the submission for publication. The Investigators in the Multi-Center (MC) study agree to postpone MC publications until the earlier of the first AstraZeneca-authorized publication or up to eighteen months from study completion at all sites.